CLINICAL TRIAL: NCT07285863
Title: An Open-Label Study On The Effects Of Human Secretin For Injection (CHIROSTIM) On Pancreatic Fluid Composition In Normal Human Volunteer Participants
Brief Title: A Study Of Effect Of Secretin For In Injection (Chirostim) On Pancreatic Fluid Composition In Healthy Subjects
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: ChiRhoClin, Inc. (Industry)
Responsible Party: Principal Investigator, Samuel Han, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25-011644
Record Dates: First submitted 2025-12-11; First posted 2025-12-16 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Exocrine Pancreatic Insufficiency; Chronic Pancreatitis
Keywords: pancreatic function test; Pancreatic fluid composition
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Pancreatitis, Chronic | interventions — Secretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Healthy Participants (Experimental): Healthy participants without pancreatic disease who are undergoing an endoscopic ultrasound for a non-pancreatic indication. This arm will be stratified into 3 age groups: 18-35, 35-45, and 46+ years. Participants will be given a standard dose of intravenous human secretin (0.2 mcg/kg) during the endoscopic ultrasound. During this time, pancreatic fluid will be collected at 5 minutes, 10 minutes, 15 minutes, and 20 minutes after secretin administration.
  Interventions: Drug: Secretin (human synthetic) - ChiRhoClin

INTERVENTIONS:
Drug: Secretin (human synthetic) - ChiRhoClin — During endoscopic ultrasound (EUS), a dose of intravenous secretin (0.2 µg/kg) will be administered over the course of 1 minute to stimulate pancreatic ductal cells to secrete pancreas fluid.
  Duodenal fluid will be aspirated through the echoendoscope in 5 minute increments (5, 10, 15, and 20 minutes) after the secretin has been administered

SUMMARY:
The purpose of this study is to collect pancreas fluid from the duodenum using the endoscopic pancreas function collection method in healthy participants after pancreatic stimulation with human secretin.

ELIGIBILITY:
Inclusion Criteria

* Males or non-pregnant females
* Age 18-80.
* Participants must be in good health based on medical history (ASA Class 3 or below)
* Participants must be willing and able to provide informed consent
* Receiving an endoscopic ultrasound for a non-pancreatic indication

Exclusion Criteria

* History of any form of pancreatitis and/or other pancreatic diseases (e.g. pancreatic cysts, pancreatic masses).
* History of inflammatory bowel disease
* History of vagotomy.
* History of surgically altered upper gastrointestinal anatomy (e.g. gastric bypass, Billroth I/II)
* History of liver disease
* Pregnant women or nursing mothers
* Regular use of anticholinergics
* > 2 drinks of alcohol daily
* Smokers (cigarette)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Pancreatic Fluid Bicarbonate Composition | 5, 10, 15, and 20-minutes post-secretin administration
  A primary outcome will be the bicarbonate level (milliequivalent per liter) in the pancreatic fluid collected.
Pancreatic Fluid Sodium Composition | 5, 10, 15, and 20-minutes post-secretin administration
  A primary outcome will be the sodium level (milliequivalent per liter) in the pancreatic fluid collected.
Pancreatic Fluid Potassium Composition | 5, 10, 15, and 20-minutes post-secretin administration
  A primary outcome will be the potassium level (milliequivalent per liter) in the pancreatic fluid collected.
Pancreatic Fluid Chloride Composition | 5, 10, 15, and 20-minutes post-secretin administration
  A primary outcome will be the chloride level (milliequivalent per liter) in the pancreatic fluid collected.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Han, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials